CLINICAL TRIAL: NCT06192745
Title: Experimental Effects of Light And Content From Evening Screen Media Use On Children's Sleep, Executive Functioning, And Emotion Regulation
Brief Title: SCREENS: Sleep, Circadian Rhythms, and Electronics in the EveNing Study
Acronym: SCREENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennette P. Moreno, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-53533; R01HD112349 (NIH)
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Sleep; Circadian Rhythm; Executive Function; Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators will be blinded to treatment condition in the analysis of outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Children will participate in 2 exposure conditions in their own homes (i.e., experimental and internal negative control), facilitated by research staff (one week apart, counterbalanced to control for possible order effects). The internal negative control will be the same for all groups, but the experimental exposure will differ. Both exposures will take place for 1 hour before bed in room lighting (40-50 lux).
  Experimental exposure: children in Group 1 will be exposed to a tablet with unfiltered bright screen light and exciting media content (BL/EC).
  Internal negative control exposure: children will participate in non-screen-based quiet activities
  Interventions: Behavioral: no screen control with dim light and calming activities; Behavioral: unfiltered Bright tablet screen; Behavioral: Exciting content
- Group 2 (Experimental): Children will participate in 2 exposure conditions in their own homes (i.e., experimental and internal negative control), facilitated by research staff (one week apart, counterbalanced to control for possible order effects). The internal negative control will be the same for all groups, but the experimental exposure will differ. Both exposures will take place for 1 hour before bed in room lighting (40-50 lux).
  Experimental exposure: children in Group 2 will be exposed to a tablet with unfiltered bright screen light and calming media content (BL/CC).
  Internal negative control exposure: children will participate in non-screen-based quiet activities
  Interventions: Behavioral: no screen control with dim light and calming activities; Behavioral: unfiltered Bright tablet screen; Behavioral: Calming Content
- Group 3 (Experimental): Children will participate in 2 exposure conditions in their own homes (i.e., experimental and internal negative control), facilitated by research staff (one week apart, counterbalanced to control for possible order effects). The internal negative control will be the same for all groups, but the experimental exposure will differ. Both exposures will take place for 1 hour before bed in room lighting (40-50 lux).
  Experimental exposure: children in Group 3 will be exposed to a tablet with filtered dim screen light and exciting media content (DL/EC).
  Internal negative control exposure: children will participate in non-screen-based quiet activities
  Interventions: Behavioral: no screen control with dim light and calming activities; Behavioral: Filtered dim tablet screen; Behavioral: Exciting content
- Group 4 (Experimental): Children will participate in 2 exposure conditions in their own homes (i.e., experimental and internal negative control), facilitated by research staff (one week apart, counterbalanced to control for possible order effects). The internal negative control will be the same for all groups, but the experimental exposure will differ. Both exposures will take place for 1 hour before bed in room lighting (40-50 lux).
  Experimental exposure: children in Group 4 will be exposed to a tablet with filtered dim screen light and calming media content (DL/CC).
  Internal negative control exposure: children will participate in non-screen-based quiet activities
  Interventions: Behavioral: no screen control with dim light and calming activities; Behavioral: Filtered dim tablet screen; Behavioral: Calming Content

INTERVENTIONS:
Behavioral: no screen control with dim light and calming activities — Non-screen-based quiet activities for 1 hour before bed in room lighting 40-50 lux
  Other Names: internal negative control
Behavioral: unfiltered Bright tablet screen — Bright light screen media exposure will be delivered on an iPad Pro provided by the research team which will be set to the brightest light intensity setting for 1 hour before bed in room lighting 40-50 lux
  Arms: Group 1; Group 2
Behavioral: Filtered dim tablet screen — Filtered dim light screen media exposure will be delivered for 1 hour before bed in room lighting 40-50 lux on an iPad Pro provided by the research team. A blue light filter will be used to alter the spectral distribution of the emitted light and the screen brightness will be dimmed to the lowest possible setting
  Arms: Group 3; Group 4
Behavioral: Exciting content — We will create a 1-hour recording of movie clips containing exciting content from age-appropriate movies for 8- to 11-year-old children as rated by Common Sense Media.
  Arms: Group 1; Group 3
Behavioral: Calming Content — We will create a 1-hour recording of movie clips containing calming content from age-appropriate movies for 8- to 11-year-old children as rated by Common Sense Media.
  Arms: Group 2; Group 4

SUMMARY:
The proposed project aims to disentangle the impact of evening light exposure emitted from tablet devices from the impact of arousing media content on children's sleep regulation, circadian physiology and next-day emotion regulation and executive functioning.

DETAILED DESCRIPTION:
Investigators will conduct a 4-group randomized, controlled trial including 200 children (8 to 11 years; Tanner stage 1 or 2) assigned to an unfiltered bright light screen (BL; 109 lux) or a dim light screen (DL; <5 lux) condition in room lighting (40-50 lux) matched with either calming (CC) or exciting content (EC). Children will participate in two weekend protocols, an experimental and a control weekend. During the experimental weekend, children will be exposed to 1 hour of tablet use in the hour before bed under the following conditions: 1) unfiltered bright screen light and exciting content (BL/EC), 2) unfiltered bright screen light and calming content (BL/CC) 3) filtered dim screen light and exciting content (DL/EC) and 4) filtered dim screen light and calming content (DL/CC). To control for the effect of screen media which is common to all 4 conditions irrespective of screen brightness and the nature of the content, each child will undergo a "control condition weekend" in which the child will participate in the same weekend study protocol, but instead of using screen media in the hour before bed, children will participate in non-screen based quiet activities in room lighting (40-50 lux). The control condition will serve as a negative internal control. The order in which children are exposed to the experimental or control weekends will be randomized (i.e., counterbalanced) to control for possible order effects.

Following a week of typical sleep and media use, a 3-day weekend protocol will be implemented in the home facilitated by research staff on two occasions (one week apart, counterbalanced). To assess a potential shift in circadian phase, dim light melatonin onset (DLMO; time at which melatonin level rise above 4pg/mL) will be assessed by research staff on Nights 1 and 3 of the weekend protocol via saliva samples collected under tightly-controlled dim light conditions (i.e., DLMO-Night 3 to DLMO-Night 1). To facilitate the assessment of circadian phases under dim light conditions (<5 lux), research staff will place temporary covers over windows and adjust the lighting in the child's bedroom. A light meter will be used to ensure appropriate lighting conditions.

On Night 2, children will be exposed to either the experimental condition to which they were assigned or the control condition. A background of room lighting (40-50 lux) will be common to both the experimental and control condition.

During the experimental condition, children will exposed to screen media according to the experimental condition they were assigned (BL/EC, BL/CC, DL/EC, DL/CC) via a handheld tablet (at eye level, 45 cm in front of the child). To standardize the distance of the iPad from the eye across participants, the tablet (or non-screen-based activity) will be placed on an adjustable bed desk at a distance of 45cm from the eye. Children will sit upright in bed with a pillow behind them. A similar posture will be used in the control condition. Assessments on Night 2, will be as follows: 1) children's sleep will be assessed via actigraphy, 2) children's arousal will be assessed via heart rate (HR), and heart rate variability (HRV) 3)subjective sleepiness ratings will be collected before the start of the experimental condition, after 30 minutes, and again at bedtime. 4) ambient light will be assessed via a light sensor clipped onto the shirt collar. The next afternoon, emotion regulation (subjective reports and respiratory sinus arrhythmia; RSA) and executive functioning (neurocognitive testing) will be measured to assess these secondary outcomes. Research staff (in teams of 2) will be present in the home to conduct the circadian phase assessments, administer the experimental conditions on the Night 2, and to conduct the executive functioning and emotion regulation assessments in the afternoon of Night 3.

During the weekend protocols, children will be able to participate in daytime activities as usual with the exception that on days when melatonin is assessed, children will be asked to refrain from strenuous physical activity as this is known to affect melatonin.

During the week prior to each weekend assessment, the procedures will be the same for all participants. Parents will select a bedtime and wake time for their child based on their habitual sleep times (+/- 30 mins). Families will be asked to maintain this sleep schedule for the duration of the 2-week protocol, except on nights when DLMO is assessed. Adherence to sleep/wake patterns will be assessed via actigraphy. Because previous exposure to light and screen media can impact future responsiveness to light and screen media, the research team will assess children's ambient light exposure using a reliable sensor clipped near the shirt collar. Mobile device screen use will be assessed using an app downloaded onto the tablet. Other types of screen media use will be assessed by parent report. Variables assessed during the weeks preceding the experimental weekend will be used as covariates in the analysis.

While 200 children are needed to be powered to examine the interaction effect of light and content on children's total sleep time, an additional 20 children will be recruited to account for attrition. The total sample size will be up 220 children.

ELIGIBILITY:
Inclusion Criteria:

* children between 8.0 and 11.9 year old
* Tanner stage 1 and 2
* live with their parent(s) (biological or legal guardian at least 50% of the time and has a primary role of caring for the child).
* Children who sleep between 8.5 to 11 hours per night habitually
* Children must sleep alone most nights
* parent and child able to communicate and read and write in English
* The child does not have to have access to a mobile device (tablet or Phone), but if they do, the primary device they use has to be an a) Android OS ≥5.0 either used only by the study child or shared with others, b) Amazon Fire OS ≥5.0 that only the child uses or c) an Apple iOS ≥14.0 that only the child uses.
* If the child's primary device is a Android or Amazon Fired device, the parent and child agree to install Chronicle App (Android or Amazon). If the child's primary device is an Apple device, the parent and child agree to allow us to gather usage screenshots from the primary iPad or iPhone.
* Families must live in the greater Houston area.

Exclusion Criteria:

* child blindness or colorblindness
* significant vision problems
* developmental or cognitive delays
* diagnosis of a sleep or psychiatric disorder
* diagnosed cognitive or learning impairment affecting executive functioning (e.g., attention deficit hyperactivity disorder)
* medical conditions that impact sleep
* taking medications that impact sleep
* travel beyond 2 time zones in the month before starting the study

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Differences in Sleep Duration on nights following the experimental and internal negative control exposures | Night 9 and 16
  Children will wear an Actiwatch Spectrum watch (Philips Respironics, Inc.) on the wrist of their non-dominant hand. Total sleep time are the total minute of sleep scored as sleep by the Sadeh algorithm between sleep onset and sleep offset.
Differences in Subjective Sleep Quality on nights following the experimental and internal negative | Night 9 and 16
  Visual analog scales will be used to collect subjective ratings of sleep quality and morning alertness the morning following the study condition. Participants will be asked to rate the quality of their sleep last night (very poor to very good), how difficult was it for them to wake up this morning (very easy to very hard), and how alert do you feel right now (wide awake to very sleepy).

SECONDARY OUTCOMES:
Differences in the change in circadian phase | night 8 to night 10 and night 15 to night 17
  Circadian phase can be examined by measuring the circadian timing of melatonin onset under dim light conditions (dim light melatonin onset; DMLO). Following established procedures with children, salivary DLMO will be collected under dim light conditions (<5 lux), via a cheek swab every 30-60 minutes beginning 5 hours prior to and ending 1-hour following typical bedtime. Saliva samples will be centrifuged, frozen, and assayed using radioimmunoassay test kits by Solid Phase in Portland Me. DLMO phase will be determined using linear interpolation across the time points before and after melatonin concentration increased to and remained above 4pg/mL. We will examine differences in the change from night 8 to night 10 and the change from night 15 to night 17.
Differences in Sleep Latency on nights following the experimental and internal negative control exposures | Night 9 and 16
  Children will wear an Actiwatch Spectrum watch (Philips Respironics, Inc.) on the wrist of their non-dominant hand. Sleep latency (i.e., the time between when they child starts to try to fall asleep as indicated by a push of the event marker button on the Actiwatch and when the child falls asleep (first 3 consecutive epochs of sleep).
Differences in Heart Rate during the experimental and internal negative exposures | Night 9 and 16
  Heart rate (HR) will be assessed using a Polar H10 HR monitor which integrates with the Actigraph GT3X-BT devices to record HR data from which raw data can be extracted. The Polar H10 HR monitor will be worn on a chest strap fitted to the child according to manufacturer guidelines during the 1-hour experimental and internal negative exposures.
Differences in Heart Rate Variability during the experimental and internal negative exposures | Night 9 and 16
  Heart rate variability (HRV) will be assessed using a Polar H10 HR monitor which integrates with the Actigraph GT3X-BT devices to record HR data from which raw data can be extracted. The Polar H10 HR monitor will be worn on a chest strap fitted to the child according to manufacturer guidelines during the 1-hour experimental and internal negative exposures.
Differences in Pre-sleep arousal scale following the the experimental and internal negative exposures | Night 9 and 16
  the Pre-Sleep Arousal Scale for Children (PSAS-C) will be used to assess Children's subjective report of arousal prior to sleep on Night 2. The PSAS-C contains 16 items comprising 2 subscales assessing somatic and cognitive arousal and demonstrated high internal consistency. Items are scored on a Likert scale from 1 to 5 with scores ranging from 16 to 80. Higher scores indicate greater pre-sleep arousal.
Differences in Subjective Sleepiness during the experimental and internal negative exposures | Night 9 and 16
  The Pictorial Sleepiness Scale is a measure of perceived sleepiness in a given moment that has been validated with individuals 4- to 73-years of age, demonstrating a strong correlation with the Karolinska Sleepiness Scale (r=.72) and the Sandford Sleepiness Scale(r=.94). The use of cartoon faces facilitates the assessment of sleepiness in population with minimal literacy skills. Almost all participants (99%) correctly ranked the faces in order of sleepiness. Children will complete the sleepiness scale before the start of the experimental condition (~60 minute prior to bedtime), 30 minutes later, and again at bedtime.
Differences in Performance on the Trier Social Stress Test following the the experimental and internal negative exposures | Day 10 and 17
  To assess objective emotion regulation in the home on Day 3, we will use a modified version the Trier Social Stress Test (TSST), The task will begin with a 5-min baseline segment, during which children will be asked to relax while they listen to a recording of nature sounds (i.e., waves at the beach) in order to collect resting HR and HRV). After this baseline period, children will then engage in a task in which they To assess objective emotion regulation in the home on Day 3, we will use a modified version the Trier Social Stress Test (TSST), The task will begin with a 5- min baseline segment, during which children will be asked to relax while they listen to a recording of nature sounds (i.e., waves at the beach) in order to collect resting HR and HRV). After this baseline period, children will then engage in a task in which they imagine they are giving a speech in front of a class of 20 kids they have never met. Resting and task-based HR and HRV data will be collected.
Differences in ratings of subjective emotion regulation following the the experimental and internal negative exposures | Day 10 and 17
  Subjective reports of emotional arousal and regulation will also be collected before and after the 5-minute speech task. Children will provide ratings of arousal using the Self-Assessment Manikin (SAM), a widely-used non-verbal pictorial scale that measures arousal associated with a person's affective reaction to a wide variety of situations and stimuli. Emotion regulation will be assessed via a likert-type rating requiring children to indicate how difficult it was to regulate (control) their emotions during the speech task, from ) (not hard at all) to 10 (very hard).
Differences in performance on the Letter Number Sequencing subtest of the WISC-V following the experimental and internal negative exposures | Day 10 and 17
  Letter-number sequencing Test (WISC-V) asks children to listen to lists of letters and digits and repeat the letters back in alphabetical order, and the digits in ascending numerical order, with the lists increasing in length from 2-8 alphanumeric characters throughout the test. Children will be read three different alphanumeric series for each list lengths, and one point will be awarded for each correct recall, for a total of 21 points. This performance score will be used as a measure of working memory.
Differences in Performance on the Delis-Kaplan Executive Function System The Color-Word Inference Test following the experimental and internal negative exposures | Day 10 and 17
  The Color-Word Interference Test (D-KEFS) is a standard "Stroop-like" task. Across the two tasks, inhibition and inhibition switching, completion time and errors (4 indicators in total) are used as markers of inhibitory control. The inhibition task is a standard "Stroop-like" task. During inhibition switching, participants also encounter words in colored ink wherein they say the color and inhibit reading the work. However, during some trials, words are enclosed by a box wherein the participant needs to switch to reading, not naming, the color in which it is printed.
Differences in Performance on the Delis-Kaplan Executive Function System The Sorting Test following the experimental and internal negative exposures | Day 10 and 17
  The Sorting Test (standard form; D-KEFS) has two conditions: free sort, and sort recognition. In free sort, children are given six cards that display both perceptual features and printed words, and asked to sort the cards into two groups, with three cards per group (description), according to as many different concepts or rules as possible (the set has a maximum of eight potential sorts), and to describe the concepts or rules as possible (the set has a maximum of eight potential sorts), and to describe the concepts employed to generate each sort, for a maximum of four minutes. In sort recognition, study staff sort the same set of cards into two groups with three cards per group, and children have a maximum of 45 seconds to identify and describe the correct sorting rule. Composite scores (based on the D-KEFS) scoring system which combines of the number of correct answers (e.g., identifying 'color' was the sort rule, with how comprehensive the description of the sort rule is.
Differences in performance on the Psychomotor Vigilance Task | Day 10 and 17
  Assesses vigilant attention (reaction time to changes in visual stimuli) and is sensitive to changes in sleep.

OTHER OUTCOMES:
Ambient Light Exposure | Days 1-17
  ActLumus devices containing a photocell will be used to assess ambient light exposure. Devices will be pinned to the shirt. ActLumus devices are capable of assessing light intensity and wavelength. Light exposure will be used as a covariate in analyses.
Average daily duration of Tablet use (excluding the experimental exposures) | Days 1-17
  Children's tablet use on Android and iOS devices will be assessed during the study period. Daily screen use will be used as a covariate in the analysis.
Other Screen Media Use | Days 1-17
  To assess for other types of screen use without over burdening parents with screen use diaries that require reporting of screen use in 15-minute increments 24 hours a day, we will add brief questions to the daily sleep diary regarding how much time (hours and minutes) the child spent on other screen devices each day (computer, video games, time spent on siblings or parent's mobile devices, t.v., etc.).
Demographics | Day 0 (baseline)
  Information will be obtained at baseline including child sex at birth and gender, parent sex and gender, parent education, family income, and child race and ethnicity. Family income-to-needs ratio will be calculated.
Structured Interviews | Screening
  Structured interviews with children and parents will be conducted at baseline over Zoom for the convenience of families. We will use the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID), a short structured diagnostic interview for assessing psychiatric disorders in children and adolescents The MINI-KID has shown excellent reliability and concordance with other validated diagnostic interview schedules for a wide range of childhood disorders. To assess for possible sleep disorders, we will conduct a brief interview with children and parents derived from the reliable B.E.A.R.S. algorithm will be used to screen for sleep problems and disorders (i.e., bed time/sleep onset problems, excessive daytime sleepiness, awakenings from sleep, regularity/duration of sleep, and snoring). Positive screens will be followed by full evaluation using diagnostic criteria for suspected sleep disorders.
Pubertal Development | Screening
  The Pubertal Development Scale (PDS) is a parent report measure consisting of five questions about pubertal status, with five answer categories (1= has not yet started changing, 2 = has barely started changing, 3 = changes are definitely underway, 4 = changes seem complete, and 0 = I do not know). A continuous PDS score is converted to a 5-point ordinal scale (in keeping with the original Tanner categories) using an algorithm described by Carskadon and Acebo. The PDS evidences high rates of test-retest reliability and agreement with clinician-performed Tanner staging.
Sleep Hygiene | Day 0 (baseline)
  Will be assessed by the Bedtime Routines Questoinnaire. The Bedtimes Routines Questionnaire (BRQ), is a 31-item parent report measure of children's bedtime routines, comprised of three scales measuring consistency of bedtime routines (weekday & weekend), reactivity to changes in bedtime routines, and frequency of adaptive and maladaptive activities. The BRQ scales had good internal consistency ranging from α = 0.69 to 0.90. Additionally, the measure has been validated in a community sample of primary caregivers of children ages 2 to 8 years old and has been used to measure bedtime routines with children ages 6 to 12 years old.
Chronotype | Day 0 (baseline)
  Chronotype refers to one's physiological preference for morningness or eveningness relative to social timing. Chronotype will be assessed during the run-in period based on parent report using the Children's Chronotype Questionnaire (CCTQ) which provides 3 measures of chronotype: 1) the midpoint of sleep on free days, 2) the morningness/Eveningness scale score, and a 5-point Chronotype score using a RedCap survey. This questionnaire has demonstrated evidence of validity to assess Chronotype among 4-11 year-olds.
Sleep Actigraphy | Days 1-7 and 11-14
  Children will wear an Actiwatch Spectrum watch (Philips Respironics, Inc.) on the wrist of their dominant hand 24-hours a day to assess sleep patterns throughout the study. This will be used to ensure that participants adhere to the bedtimes and waketimes recommended in the study protocol. Actigraphy is a reliable method for determining sleep-wake patterns in children. The Actiwatch Spectrum is a lightweight watch that collects continuous movement data in 1-minute epochs via a highly sensitive piezo-electric accelerometer. Children (with reminders from caregivers) press a button on the watch each day when they get into bed and when they get out of bed (i.e., event markers) to provide a reliable estimation of the nighttime sleep period. The watch also has an off-wrist sensor which beeps to remind the child to put on the watch when taken off. The validated Sadeh algorithm will be used to derive the bed time and wake time to examine adherence to the sleep schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Jennette P Moreno, PhD, Principal Investigator — Baylor College of Medicine; Candice A Alfano, PhD, Principal Investigator — University of Houston
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the National Institute of Child Health and Human Development-maintained Data and Specimen Hub (DASH) data repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available for a minimum of 3 years following the closeout of the grant, though data will be retained at Baylor College of Medicine for a minimum of 7 years following the close-out of the study.
Access Criteria: Access to the data will be controlled by the repository.